CLINICAL TRIAL: NCT06878300
Title: Assessing Functional Outcomes and User Experience of the Lexie B3 Pro Powered by Bose Over-the-counter Self-Fitting Hearing Aid in Adults With Perceived Mild-Moderate Hearing Loss: A Three Phased Approach
Brief Title: Assessing Functional Outcomes and User Experience of the Lexie B3 Pro Powered by Bose Over-the-counter Self-Fitting Hearing Aid
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn before enrollment for administrative reasons.
Sponsor: HearX SA (Industry)
Responsible Party: Sponsor
Organization: hearX Group (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LexieB3Pro
Record Dates: First submitted 2025-03-11; First posted 2025-03-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss; Self Perceived Hearing Loss; Hearing Impairment
Keywords: over the counter hearing aids; self-fitting hearing aids; hearing aids
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTC SF (Lexie) (Experimental): Participants in this group will be provided with a Lexie self-fitting OTC hearing aid that features a proprietary fitting algorithm designed to optimize amplification settings based on user input. Participants will independently set up and adjust the device without professional assistance, following the manufacturer's instructions, as would be the standard use case for self-fitting hearing aids. They will use the device for a two-week take-home field trial before crossing over to the alternative study arm.
  Interventions: Device: Over the counter hearing aid (Lexie)
- OTC SF Competitor (Experimental): Participants in this group will receive a different self-fitting OTC hearing aid that utilizes its own manufacturer-specific fitting approach. As in the experimental arm, participants will complete the setup independently without professional guidance, adjusting the device based on the available self-fitting process. They will use this device for a two-week take-home field trial before switching to the experimental arm.
  Interventions: Device: Comparator over the counter hearing aid

INTERVENTIONS:
Device: Over the counter hearing aid (Lexie) — The study will compare user perceptions of two over-the-counter (OTC) hearing aids, with the Lexie B3 Pro serving as the reference device. Participants will be fitted with each device for a predetermined period in a randomized order to ensure balanced exposure.
  Arms: OTC SF (Lexie)
Device: Comparator over the counter hearing aid — The comparator OTC hearing aid will undergo the same evaluation process as the Lexie B3 Pro, ensuring an equivalent and unbiased comparison. Participants will be provided with the comparator device along with its standard user instructions, including any mobile applications or self-fitting guidance designed for independent setup.
  Arms: OTC SF Competitor

SUMMARY:
Hearing loss significantly impacts quality of life, with sensorineural hearing loss being the most common type among adults. Hearing aids are a well-established intervention, yet barriers such as access and affordability limit their adoption, even in countries with developed audiological services . Despite their proven benefits, many individuals who could benefit from hearing aids do not obtain them. Traditionally, hearing aids required professional consultations, which created access challenges. In 2022, the U.S. FDA approved over-the-counter (OTC) hearing aids, including self-fitting devices, to improve accessibility. Recent clinical trials suggest that OTC hearing aids can provide similar benefits to professionally fitted ones in speech recognition and self-reported outcomes.

One critique of past studies is that they often compare OTC hearing aids to audiologist-fitted devices using the same hardware, with differences primarily in programming methods. While much research has focused on fitting methods, this study aims to evaluate a new OTC hearing aid with its proprietary fitting algorithm against a marketed competitor. This randomized controlled trial (RCT) forms part of a larger validation study that follows a phased approach. Phase 1 validates an in-situ hearing test against a standard audiometer and Phase 2 assesses user experience. This RCT (Phase 3) will compare two OTC devices-the Lexie B3 Pro and a competitor already on the market-to evaluate self-reported benefit, user experience, and satisfaction. The hypothesis is that both devices provide comparable outcomes.

DETAILED DESCRIPTION:
Hearing loss is a prevalent global health concern with significant social, emotional, and economic consequences. Sensorineural hearing loss (SNHL) is the most common type among adults, often resulting from aging, noise exposure, or ototoxic medication. Left untreated, hearing loss can lead to communication difficulties, social isolation, depression, cognitive decline, and reduced quality of life. Hearing aids are the most widely used intervention for addressing hearing impairment, offering substantial benefits in speech perception, communication, and overall well-being. However, despite the well-documented advantages of hearing aids, adoption rates remain low across various populations.

Barriers to hearing aid adoption include cost, accessibility, stigma, and the traditional requirement for professional fitting. In many countries, hearing aids are expensive, and access to hearing healthcare professionals is limited, particularly in rural or underserved areas. Even in regions with well-established audiological services, individuals may face challenges such as lengthy appointment wait times, insurance limitations, or the perception that hearing aids are not necessary until hearing loss is severe.

To address accessibility challenges, the U.S. Food and Drug Administration (FDA) introduced regulations in 2022 allowing the sale of over-the-counter (OTC) hearing aids. These devices are designed for adults with perceived mild-to-moderate hearing loss and can be purchased without the need for a professional hearing assessment or fitting. OTC hearing aids aim to lower barriers by providing a more affordable, convenient, and consumer-driven option. Among OTC hearing aids, self-fitting models offer additional benefits, as users can fine-tune their settings using built-in hearing tests or app-based adjustments, potentially achieving outcomes comparable to those of audiologist-fitted hearing aids.

Emerging research suggests that OTC hearing aids can be effective in improving speech recognition and self-reported hearing outcomes, with some studies indicating that self-fitting devices perform similarly to traditional, professionally fitted hearing aids. However, there is ongoing debate regarding the best methods for fitting and personalizing these devices. Previous research has often compared OTC hearing aid fitting methods to audiologist fittings using the same hardware, with the primary difference being the programming approach rather than the device itself. This approach has drawn criticism because it does not fully reflect real-world consumer decisions, where individuals must choose between different OTC models with varying features, fitting algorithms, and user interfaces.

This study aims to address this gap by directly comparing two distinct OTC hearing aids: the Lexie B3 Pro, which features a proprietary self-fitting algorithm, and a competing marketed device. The goal is to assess whether both devices offer comparable outcomes in terms of self-reported benefit, user experience, and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be 18 years or older.
* The outer ear must be free from excessive cerumen, outer or middle ear disease.
* The participant must have bilateral self-perceived mild-moderate hearing loss.
* Baseline pure tone evaluations should fall within a 4-frequency PTA (0.5, 1.0, 2.0, 4.0 kHz) of 65 dB HL or less.
* The participant must have an adequate level of English proficiency as measured objectively using an English proficiency test (EF SET).
* The participant must present with Type A or As or Ad tympanogram as measured by tympanometry.
* Must be in possession of a smartphone compatible with the Lexie App (Android OS 8)

Exclusion Criteria:

* Younger than 18 years
* Severe or greater hearing loss
* Outer or middle ear abnormality
* Have any of the following as per FDA (21 CFR 801.420) reg-flag conditions as contraindications to OTC hearing aid use :

  (i) Visible congenital or traumatic deformity of the ear preventing insertion of the receiver wire and dome into the ear.

(ii) History of sudden active drainage (i.e. blood or pus) from the ear within the previous 6 months.

(iii) Painful or uncomfortable feeling in your ear (iv) Visible evidence of significant cerumen accumulation or a foreign body in the ear canal.

(v) History of sudden or rapidly progressive hearing loss within the previous 6 months.

(vi) Acute or chronic dizziness. (vii) Unilateral hearing loss. (viii) Fluctuating hearing loss (ix) Unilateral tinnitus

* Low English proficiency - <51% of EF-SET
* No access or in possession of an Android smartphone, compatible with the Lexie App (minimum Android OS 8)

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Hearing aid perception questionnaire | At the end of the two week field trial (with each device)
  To achieve the study's primary objective of comparing the self-fitting Lexie B3 Pro OTC hearing aid device with the comparable market-available OTC self-fitting device, the primary outcome will be measured using a self-developed questionnaire with Likert scale questions. This questionnaire is designed to gather detailed insights into participants' perceptions of the devices' features and their experiences using both the self-fitting Lexie B3 Pro device and the market-available model after completing each field trial. No specific scoring is used as the study aims to obtain descriptive insights between the two devices.

CONTACTS AND LOCATIONS:
Overall Officials: Karina C De Sousa, PhD, Principal Investigator — hearX Group

IPD SHARING:
Plan to Share IPD: No
The study is conducted under the South African Health Products Regulatory Authority (SAHPRA) and US Food and Drug Administration (FDA) Institutional regulations, which impose strict guidelines on the handling and sharing of medical device trial data. Furthermore, the data may contain proprietary or commercially sensitive information related to the device's performance. Sharing IPD could compromise intellectual property or competitive interests of the device manufacturer. While the raw IPD will not be shared, aggregate-level data, summary statistics, and study findings may be published and made available in peer-reviewed journals and reports.